CLINICAL TRIAL: NCT05240300
Title: A Phase 1b/2a, Double-blind (Sponsor Open), Randomized, Vehicle-controlled Study of Topically Administered BX005-A in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Topical BX005-A in Subjects With Moderate to Severe Atopic Dermatitis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study did not start enrollment due to business reasons
Sponsor: BiomX, Inc. (Industry)
Collaborators: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMX-05-001
Record Dates: First submitted 2022-01-23; First posted 2022-02-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BX005-A (Experimental): twice daily topical application x 8 weeks
  Interventions: Biological: BX005-A
- Vehicle (Placebo Comparator): twice daily topical application x 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BX005-A — phage gel
  Arms: BX005-A
Other: Placebo — vehicle gel
  Arms: Vehicle

SUMMARY:
The purpose of study BMX-05-001 is to evaluate the safety, tolerability, efficacy, and pharmacodynamics of BX005-A compared to vehicle administered topically in adult subjects with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
BMX-05-001 is a double-blind (Sponsor open), randomized, vehicle-controlled, first-in-human, Phase 1b/2a study to evaluate the safety, tolerability, efficacy, and pharmacodynamics of BX005-A compared to vehicle administered topically twice daily for 8 weeks to lesional areas in adult subjects with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old
2. Confirmed clinical diagnosis of active AD with at least a 6-month history and clinically stable AD for ≥ 1 month
3. Clinical diagnosis of moderate or severe AD with a vIGA-AD score of ≥ 3 and a lesion vIGA-AD score ≥ 3 in the target AD skin lesion
4. BSA with AD of 2%-30%, excluding scalp
5. Colonized with S. aureus in at least one AD skin lesion
6. Female subjects of non-childbearing potential must meet at least 1 of the following: postmenopausal status; documented hysterectomy and/or bilateral oophorectomy; or medically confirmed ovarian failure. All other female subjects (including those who have undergone tubal ligation) are of childbearing potential.
7. Female subjects of childbearing potential who have a negative urine pregnancy test
8. Effective contraceptive method for female subjects of childbearing potential and for male subjects
9. Able to understand study procedures and attend all study visits
10. Willing to refrain from use of all other systemic or topical agents for the treatment of AD or the prevention of complications of AD (e.g., secondary infection)

Exclusion Criteria:

1. Active skin infection and/or systemic infection requiring systemic or topical antimicrobial agents and/or a skin drainage procedure, or a history of recurrent bacterial skin infections
2. Other concurrent skin diseases which could interfere with the diagnosis and/or management of AD (e.g., psoriasis, contact dermatitis), or presence of open, chronic non-healing wounds in their treatable AD lesions
3. Known hypersensitivity to study drug, its excipients, simethicone, and/or any emollient to be used in study
4. Planned treatment with a prohibited medication during study, or received a prohibited medication within time frame noted below, prior to first dose of study drug:

   Must be discontinued at least 28 Days prior to Day 1:
   * Systemic corticosteroids
   * Systemic JAK inhibitors and immunosuppressive agents
   * Nonbiologic investigational agent or device
   * Total body phototherapy

   Must be discontinued at least 14 Days prior to Day 1:
   * Systemic antimicrobials
   * Probiotics and prebiotics
   * Prescription skin barrier repair products

   Must be discontinued at least 7 Days prior to Day 1:
   * Topical therapies for AD
   * Topical antimicrobials and antiseptic cleansers
   * Use of antibacterial soaps or topical sodium hypochlorite-based products
   * Current emollient use (need to convert to study emollient 7 days prior to Day 1)
5. Currently being treated with biologic agents; exception: may be enrolled if dupilumab was discontinued at least 12 weeks prior to Day 1, or if other biologics were discontinued at least 5 half-lives prior to Day 1.
6. Female subjects who are pregnant, breastfeeding, or planning a pregnancy, or are of childbearing potential and not using an effective and allowed form of contraception.
7. Enrolled in another investigational study 30 days prior to Screening or 90 days prior to Screening if investigational agent was a phage product.
8. Other medical and/or psychiatric conditions which makes the subject inappropriate for study participation, increases likelihood that the subject will not be able to comply with study therapy or procedures and/or which places the subject at undue risk
9. Active abuse of alcohol and/or illicit drugs or a history of such abuse that would make it difficult for the subject to comply with study and/or place subject at undue risk
10. Known infection with human immunodeficiency virus (HIV) or other immunodeficiency disorder.
11. Current or prior history of a malignant neoplasm other than previously treated non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: adverse events (AEs) | Through study completion Day 225 (+7 days)
  The proportion of subjects with any AE, treatment-emergent AE (TEAE), serious adverse event, TEAE leading to study drug discontinuation, TEAE leading to study discontinuation, or death
Safety and tolerability: laboratory abnormalities | Through study completion Day 225 (+7 days)
  The proportion of subjects with abnormalities in laboratory parameters, graded according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials

SECONDARY OUTCOMES:
Change from baseline in log S. aureus density, measured by colony forming units (CFU)/cm2 in the target AD skin lesion in BX005-A vs vehicle groups | Day 1 through Day 71 (± 2 days)
  S. aureus CFU in target AD skin lesion
Change from baseline in log S. aureus density, measured by quantitative PCR (qPCR)/cm2 in the target AD skin lesion in BX005-A vs vehicle groups | Day 1 through Day 71 (± 2 days)
  S. aureus qPCR in target AD skin lesion
% change from baseline in the Eczema Area and Severity Index (EASI) score in BX005-A vs vehicle groups | Day 1 through Day 71 (± 2 days)
  Eczema Area and Severity Index of all lesional skin areas (range 0-72); higher score indicates worse atopic dermatitis
Proportion of subjects who achieve a Validated Investigator Global Assessment AD (vIGA-AD) score of 0 or 1 with at least a 2-grade reduction from baseline in BX005-A vs vehicle groups | Day 1 through Day 71 (± 2 days)
  vIGA-AD
Change from baseline in SCORing Atopic Dermatitis (SCORAD) index in BX005-A vs vehicle groups | Day 1 through Day 71 (± 2 days)
  SCORing Atopic Dermatitis index of all lesional skin areas (range 0-103); higher score indicates worse atopic dermatitis
Change from baseline in SCORing Atopic Dermatitis (SCORAD) index of the target AD skin lesion in BX005-A vs vehicle groups | Day 1 through Day 71 (± 2 days)
  Local SCORing Atopic Dermatitis index (range 0-15); higher score indicates worse atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, Study Director — BiomX, Inc.

IPD SHARING:
Plan to Share IPD: No